CLINICAL TRIAL: NCT07298395
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 12-Week Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ENV 294 in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of ENV-294 in Adults With Moderate-to-Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Enveda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENV-294-201
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENV-294 Treatment Arm (Experimental): ENV-294 will be administered to those participants randomized to the treatment arm.
  Interventions: Drug: ENV-294
- Placebo Arm (Placebo Comparator): A placebo (matching the appearance of the experimental drug) will be administered to those participants who are randomized to the placebo arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENV-294 — ENV-294 is an orally administered investigational drug supplied as capsules. Each participant will receive ENV-294 at a total dose of 800 milligrams (mg) once daily by mouth for 12 weeks. Capsules should be taken with water, approximately the same time each day, with or without food, as directed by the study physician.
  Arms: ENV-294 Treatment Arm
Drug: Placebo — Matching oral capsule that does not contain active drug. Administered once daily by mouth for 12 weeks under the same conditions as the investigational product.
  Arms: Placebo Arm

SUMMARY:
The goal of this clinical trial is to learn about the safety and effectiveness of ENV-294 in adults with moderate to severe atopic dermatitis.

The main questions it will answer are:

* Is there an impact on the severity and area of atopic dermatitis when participants take ENV-294
* What medical problems do participants have when taking ENV-294 Researchers will review the atopic dermatitis present at the beginning of the study against the atopic dermatitis present at the end of the study.

Participants will:

* Take drug ENV-294 or a placebo once every day for 12 weeks
* Visit the clinic every 2 to 4 weeks for checkups and tests
* Keep a diary of their symptoms and when they took their study drug ENV-294
* Return to the clinic for the final study visit at approximately week 16

ELIGIBILITY:
Inclusion Criteria:

* Have chronic atopic dermatitis that was diagnosed at least 12 months prior to the first study visit
* Have had either: (1) a poor response or intolerance to topical treatments for atopic dermatitis (such as corticosteroids) within the past 6 months, as determined by the study doctor, or (2) a poor response to treatments administered by mouth within the past 12 months.
* Use a bland moisturizer at least daily

Exclusion Criteria:

* Current or recurrent medical conditions that could affect the study drug or study assessments, including but not limited to: cardiovascular, neurological, kidney, liver, gastrointestinal, cancer, autoimmune disease, HIV, hepatitis B, hepatitis C, or psychiatric disorders.
* Any illness that could impact participant safety, clinically significant depression (as determined by the investigator), or active bacterial, fungal, or viral infections.
* Have an ongoing skin condition or large tattoos that would interfere with the clinical assessment, evaluation of atopic dermatitis, or treatment response.
* Have an ongoing clinically significant skin infection or receiving treatment for infection that may interfere with assessment of atopic dermatitis.
* Have clinically significant abnormal clinical laboratory assessments at the first or second study visit as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of ENV-294 compared to placebo on severity and extent of atopic dermatitis (AD) | Baseline to Week 12 (Day 85)
  The effectiveness of ENV-294 compared with placebo will be assessed by the percent change in Eczema Area and Severity Index (EASI) score from the start of the study (Baseline) to Week 12 (Day 85). The EASI score measures the extent and severity of atopic dermatitis, with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events | Baseline to Week 12 (Day 85)
  1. Number and seriousness of adverse events (AEs), serious adverse events (SAEs), and adverse events leading to discontinuation of study drug.
To evaluate how well ENV-294 works in participants with atopic dermatitis during 12 weeks of treatment. | Baseline to Week 12 (Day 85)
  1. Percentage of participants with at least 75% reduction from Baseline in Eczema Area and Severity Index (EASI) score at Week 12.
To evaluate pharmacokinetics (PK) using limited blood samples during the 12-week treatment period. | Baseline through Week 12 (Day 85)
  Observed concentration values of ENV-294 at the times blood samples are collected during the 12-week treatment period.
Observed values, change from baseline, and percent change from baseline in heart rate (beats per minute) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the end of study at approximately week 16.
  Heart rate measured from 12-lead ECG recordings in beats per minute to assess cardiac safety and tolerability.
Observed value, change from baseline, and percent change from baseline in systolic blood pressure (mmHg) as a measure of safety and tolerability. | Baseline through the end of the treatment period and the end of the study at approximately week16.
  Systolic blood pressure measured in millimeters of mercury (mmHg) using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294..
To assess the efficacy of ENV-294 in participants with AD over a 12- Week treatment period | Baseline through Week 12
  Proportion of participants who achieve a ≥2-point reduction from Baseline in Validated Global Investigator Assessment (vIGA) score and a score of 0 or 1 at Week 12
To evaluate how well ENV-294 works in participants with atopic dermatitis during 12 weeks of treatment. | Baseline through Week 12
  Change and percent change in Patient Oriented Eczema Measure (POEM) at Week 12
To evaluate how well ENV-294 works in participants with atopic dermatitis during 12 weeks of treatment. | Baseline through Week 12
  Peak Pruritus Numerical Rating Scale (PP-NRS) response status defined as achieving weekly mean decreases of ≥4 points
Observed value, change from baseline, and percent change from baseline in diastolic blood pressure (mmHg) as a measure of safety and tolerability. | Baseline through the end of the treatment period at approximately week 16.
  Diastolic blood pressure measured in millimeters of mercury (mmHg) using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294
Observed value, change from baseline, and percent change from baseline in heart rate (beats per minute) as a measure of safety and tolerability. | Baseline throug the treatment period and the end of study at approximately week 16.
  Heart rate measured in beats per minute (bpm) using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Observed value, change from baseline, and percent change from baseline in respiratory rate (breaths per minute) as a measure of safety and tolerability. | Baseline through the treatment priod and the end of the study at approximately week 16
  Respiratory rate measured in breaths per minute using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Observed values, change from baseline, and percent change from baseline in RR interval (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  RR interval measured from 12-lead ECGs in milliseconds (ms) to assess cardiac safety and tolerability.
Observed values, change from baseline, and percent change from baseline in PR interval (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  PR interval measured in milliseconds (ms) using standard 12-lead ECGs to assess safety and tolerability.
Observed values, change from baseline, and percent change from baseline in QRS duration (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QRS duration measured in milliseconds (ms) using standard 12-lead ECGs to assess cardiac conduction and safety.
Observed values, change from baseline, and percent change from baseline in QT interval (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QT interval measured in milliseconds (ms) using standard 12-lead ECGs to assess cardiac repolarization safety.
Observed values, change from baseline, and percent change from baseline in QTc Bazett (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QTc Bazett (QT corrected for heart rate using Bazett's formula) measured in milliseconds (ms) to evaluate cardiac safety.
Observed values, change from baseline, and percent change from baseline in QTc Fridericia (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QTc Fridericia (QT corrected for heart rate using Fridericia's formula) measured in milliseconds (ms) to evaluate cardiac safety.

CONTACTS AND LOCATIONS:
Overall Officials: Gurpreet Ahluwalia, PhD, Study Director — Enveda Therapeutics
Locations (1):
- Options Research Group, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The data include sensitive health information that cannot be fully de-identified under current privacy standards, and the sponsor does not plan to make IPD available outside the study team. Summary results and aggregate data will be shared publicly as required by regulation.